CLINICAL TRIAL: NCT00109590
Title: Phase II Study of the Pharmacokinetics of Nevirapine and the Incidence of Nevirapine Resistance Mutations in HIV-Infected Women Receiving a Single Intrapartum Dose of Nevirapine With the Concomitant Administration of Zidovudine/Didanosine or Zidovudine/Didanosine/Lopinavir/Ritonavir
Brief Title: Reducing the Incidence of Nevirapine Resistance Mutations in Pregnant HIV Infected Women Who Receive Anti-HIV Drugs Prior to and After Giving Birth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1032; 10137 (Registry Identifier: DAIDS ES); PACTG P1032
Record Dates: First submitted 2005-04-29; First posted 2005-05-02 (Estimated); Results first posted 2012-11-06 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2019-01

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; Treatment Naive; Pregnancy; Perinatal Transmission; Vertical Transmission; Mother-To-Child Transmission; MTCT
MeSH Terms: conditions — HIV Infections | interventions — Didanosine; Lopinavir; Nevirapine; Zidovudine

ARMS (3):
- Arm A: LPV/r x 7d (Experimental): NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, every 3 hours during labor and BID for 7 days postpartum, ddI 250 mg orally daily (if body weight <60 kg) or 400 mg orally twice daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 7 days postpartum, LPV/r 400/100mg orally twice daily at the onset of labor, during labor and for 7 days postpartum.
  Interventions: Drug: Didanosine, enteric-coated; Drug: Lopinavir/ritonavir; Drug: Nevirapine; Drug: Zidovudine
- Arm B: no LPV/r (Experimental): NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, every 3 hours during labor and twice daily for 7 days postpartum , ddI 250 mg orally daily (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 30 days postpartum.
  Interventions: Drug: Didanosine, enteric-coated; Drug: Nevirapine; Drug: Zidovudine
- Arm C: LPV/r x 30d (Experimental): NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, every 3 hours during labor and twice daily for 7 days postpartum , ddI 250 mg orally daily (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 30 days postpartum,LPV/r 400/100mg orally twice daily at the onset of labor, during labor and for 30 days postpartum.
  Interventions: Drug: Didanosine, enteric-coated; Drug: Lopinavir/ritonavir; Drug: Nevirapine; Drug: Zidovudine

INTERVENTIONS:
Drug: Didanosine, enteric-coated — once daily
Drug: Lopinavir/ritonavir — twice daily
  Arms: Arm A: LPV/r x 7d; Arm C: LPV/r x 30d
Drug: Nevirapine — single-dose at the onset of labor
Drug: Zidovudine — twice daily

SUMMARY:
The purpose of this study is to determine which of 3 different anti-HIV drug regimens given to HIV infected pregnant women during and after their pregnancies is most effective in reducing the incidence of nevirapine (NVP) resistance mutations. Blood levels of NVP and lopinavir/ritonavir (LPV/r) will also be studied.

Study hypothesis: NVP resistance following single-dose NVP can be prevented with the concomitant administration of additional antiretroviral therapy (ART).

DETAILED DESCRIPTION:
A single dose of nevirapine (SD-NVP) given to an HIV infected pregnant woman in labor followed by a single dose to her infant had been shown to be a simple and effective means of reducing mother-to-child transmission (MTCT) of HIV among women who had not received antiretroviral (ART) during pregnancy. However, development of NVP and other nonnucleoside reverse transcriptase inhibitor (NNRTI)-resistant virus was a concern. An optimal ART regimen that can prevent selection of resistant virus while efficiently preventing MTCT was needed. This study evaluated 3 different ART strategies for preventing the development of NVP resistance in HIV infected pregnant women and compared the incidence of NVP resistance mutations postpartum observed with each regimen to the incidence among historical controls. NVP and LPV/r pharmacokinetics (PK) were also evaluated in this study.

Participants were randomly assigned to one of three study arms. All study participants received a single dose of oral NVP at the onset of labor and, oral zidovudine (ZDV) at the onset of labor, and every three hours during labor. Arm A: (LPV/r x 7d) participants received enteric-coated didanosine (ddI) and LPV/r orally twice daily beginning at the onset of labor and continuing through 7 days postpartum; oral ZDV was also taken twice daily for 7 days postpartum. Arm B: (no LPV/r) participants received enteric-coated ddI beginning at the onset of labor and continued through 30 days postpartum; oral ZDV was also taken twice daily for 30 days postpartum. Arm C : (LPV/r x 30d) participants received enteric-coated ddI and LPV/r orally twice daily beginning at the onset of labor and continued through 30 days postpartum; oral ZDV was also taken twice daily for 30 days postpartum.

All women were followed for at least 24 weeks postpartum. Women with resistance mutations identified within 8 weeks postpartum were to be followed until 72 weeks postpartum to evaluate the persistence of the mutations. All infants were followed until at least 12 weeks of age. HIV-infected infants were to be followed until 24 weeks of age. There were 11 study visits for women at day 10, 21, and 30 and week 5, 6, 8, 12, 24, 36, 48, and 72. Medical history assessment, a physical exam, and blood collection occurred at all visits. Blood collection for PK studies occurred at Days 10, 21, and 30. All women were asked to complete an adherence questionnaire at Day 10; women assigned to Arms A : LPV/r x 7d and B: no LPV/r were also asked to complete an adherence questionnaire at Day 30. There were 6 study visits for infants at birth - 48 hours, day 21, week 5, 12, 16 and 24. Medical history assessment and a physical exam occurred at most visits; blood collection occurred at all visits.

Data and specimens for the historical control comparison group were obtained from the PHPT-2 trial*, in which five of the P1032 study sites had participated between 2001 and 2003. PHPT-2 was a study of the efficacy of SD-NVP to prevent MTCT among women who received ZDV after 27 weeks gestation but no postpartum ART. Criteria for inclusion in the historical comparison group included receipt of SD-NVP, a CD4 count of more than 250 cells per cubic millimeter within 30 days of screening or entry, and the availability of plasma samples at 10 days or 6 weeks post-partum.

* Lallement M, Jourdain G, Le Coeur S, et al. Single-dose perinatal nevirapine plus standard zidovudine to prevent mother-to-child transmission of HIV-1 in Thailand. N Engl J Med 2004; 351:217-28.

ELIGIBILITY:
Inclusion Criteria for Mothers:

* HIV infected
* Pregnant with a viable fetus
* Between 28 and 38 weeks of pregnancy
* CD4 count greater than 250 cells/mm3 within 30 days prior to study entry
* Able to receive oral ART during labor
* Willing to use acceptable forms of contraception while on study treatment
* Able to provide written informed consent

Exclusion Criteria for Mothers:

* Known allergy or hypersensitivity to ddI, LPV, NVP, ritonavir (RTV), or ZDV
* Any ART other than ZDV during a previous pregnancy or the current pregnancy
* Certain medications
* Planning to receive additional ART during the first 8 weeks postpartum
* Planning to breastfeed
* Unlikely to comply with postpartum study requirements, in the opinion of the investigator
* Certain abnormal laboratory values within 30 days prior to study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2006-06; Primary Completion 2008-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Van Dyke, MD, Study Chair — Tulane University Medical School; Gonzague J. Jourdain, MD, Study Chair — Program for HIV Prevention and Treatment / IRD054, Department of Immunology and Infectious Diseases, Harvard School of Public Health
Locations (7):
- Thailand (7):
  - Bhumibol Adulyadej Hosp. CRS, Saimai, Bangkok
  - Siriraj Hospital Mahidol University CRS, Bangkok, Bangkoknoi
  - Prapokklao Hosp. CRS, Chanthaburi
  - Chiang Mai University Pediatrics-Obstetrics CRS, Chiang Mai
  - Chiangrai Prachanukroh Hospital CRS, Chiangrai
  - Chonburi Hosp. CRS, Chon Buri
  - Phayao Provincial Hosp. CRS, Phayao

REFERENCES:
- [Background] Cunningham CK, Chaix ML, Rekacewicz C, Britto P, Rouzioux C, Gelber RD, Dorenbaum A, Delfraissy JF, Bazin B, Mofenson L, Sullivan JL. Development of resistance mutations in women receiving standard antiretroviral therapy who received intrapartum nevirapine to prevent perinatal human immunodeficiency virus type 1 transmission: a substudy of pediatric AIDS clinical trials group protocol 316. J Infect Dis. 2002 Jul 15;186(2):181-8. doi: 10.1086/341300. Epub 2002 Jun 26. PMID 12134253
- [Background] Lyons FE, Coughlan S, Byrne CM, Hopkins SM, Hall WW, Mulcahy FM. Emergence of antiretroviral resistance in HIV-positive women receiving combination antiretroviral therapy in pregnancy. AIDS. 2005 Jan 3;19(1):63-7. doi: 10.1097/00002030-200501030-00007. PMID 15627034
- [Background] Sullivan JL. Prevention of mother-to-child transmission of HIV--what next? J Acquir Immune Defic Syndr. 2003 Sep;34 Suppl 1:S67-72. doi: 10.1097/00126334-200309011-00010. PMID 14562860
- [Background] Thorne C, Newell ML. The safety of antiretroviral drugs in pregnancy. Expert Opin Drug Saf. 2005 Mar;4(2):323-35. doi: 10.1517/14740338.4.2.323. PMID 15794723
- [Result] Cressey TR, Van Dyke R, Jourdain G, Puthanakit T, Roongpisuthipong A, Achalapong J, Yuthavisuthi P, Prommas S, Chotivanich N, Maupin R, Smith E, Shapiro DE, Mirochnick M; IMPAACT P1032 Team. Early postpartum pharmacokinetics of lopinavir initiated intrapartum in Thai women. Antimicrob Agents Chemother. 2009 May;53(5):2189-91. doi: 10.1128/AAC.01091-08. Epub 2009 Feb 23. PMID 19237646
- [Result] Van Dyke RB, Ngo-Giang-Huong N, Shapiro DE, Frenkel L, Britto P, Roongpisuthipong A, Beck IA, Yuthavisuthi P, Prommas S, Puthanakit T, Achalapong J, Chotivanich N, Rasri W, Cressey TR, Maupin R, Mirochnick M, Jourdain G; IMPAACT P1032 Protocol Team. A comparison of 3 regimens to prevent nevirapine resistance mutations in HIV-infected pregnant women receiving a single intrapartum dose of nevirapine. Clin Infect Dis. 2012 Jan 15;54(2):285-93. doi: 10.1093/cid/cir798. Epub 2011 Dec 5. PMID 22144539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled at seven IMPAACT affiliated sites in Thailand. Between June 9, 2006 and June 30, 2008, 175 participants enrolled in the study.
Pre-assignment Details: The study recruited HIV infected pregnant women who were >= 18 years of age,>=28 to <38 weeks gestation, who did not plan to start antiretroviral treatment within eight weeks following delivery, not planning to breastfeed and had CD4+ count >250 cells/mm3. Women were randomized in approximately equal numbers to one of three treatment arms.
Groups:
- Arm A : LPV/r x 7d: Nevirapine (NVP) 200 mg orally, single dose at onset of labor, Zidovudine (ZDV) 300 mg orally at onset of labor, every 3 hours during labor and twice daily for 7 days postpartum, didanosine (ddI) 250 mg orally (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 7 days postpartum,> Lopinavir/Ritonavir (LPV/r) 400/100mg orally twice daily at the onset of labor, during labor and for 7 days postpartum.
- Arm B : no LPV/r: Neviarpine (NVP) 200 mg orally, single dose at onset of labor, Zidovudine (ZDV) 300 mg orally at onset of labor, every 3 hours during labor and twice daily for 30 days postpartum, didanosine (ddI) 250 mg orally (if body weight <60 kg) or 400 mg orally once daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 30 days postpartum.
- Arm C: LPV/r x 30d: Nevirapine (NVP) 200 mg orally, single dose at onset of labor, Zidovudine (ZDV) 300 mg orally at onset of labor, every 3 hours during labor and twice daily for 30 days postpartum, didanosine (ddI) 250 mg orally (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 30 days postpartum, Lopinavir/Ritonavir (LPV/r) 400/100mg orally twice daily at the onset of labor, during labor and for 30 days postpartum.
Period: Overall Study
Arm/Group | Arm A : LPV/r x 7d | Arm B : no LPV/r | Arm C: LPV/r x 30d
Started | 57 | 58 | 60
RECEIVED TREATMENT | 56 | 56 | 57
Completed | 55 | 56 | 56
Not Completed | 2 | 2 | 4
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Never Started Treatment | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Arm A : LPV/r x 7d: NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, every 3 hours during labor and twice daily for 7 days postpartum, ddI 250 mg orally (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 7 days postpartum, LPV/r 400/100mg orally twice daily at the onset of labor, during labor and for 7 days postpartum.
- Arm B : no LPV/r: NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, every 3 hours during labor and twice daily for 30 days postpartum, ddI 250 mg orally (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 30 days postpartum.
- Arm C: LPV/r x 30d: NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, evry 3 hours during labor and twice daily for 30 days postpartum, ddI 250 mg orally (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 30 days postpartum, LPV/r 400/100mg orally twice daily at the onset of labor, during labor and for 30 days postpartum.
- Total: Total of all reporting groups
Arm/Group | Arm A : LPV/r x 7d | Arm B : no LPV/r | Arm C: LPV/r x 30d | Total
Number analyzed (Participants) | 56 | 56 | 57 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (6) | 28 (5) | 27 (5) | 28 (5)
Age, Customized [Number; unit: participants]
  18 to < 30years | 34 | 35 | 38 | 107
  >=30 to < 45 years | 21 | 21 | 19 | 61
  >= 45 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 56 | 57 | 169
  Male | 0 | 0 | 0 | 0
Gestational Age at Entry [Median (Full Range); unit: weeks] | 32 [28 to 37] | 31 [27 to 38] | 31 [28 to 37] | 31 [27 to 38]
Duration of ZDV during pregnancy - At Entry [Median (Full Range); unit: weeks] | 3 [0 to 9] | 2 [0 to 10] | 2 [0 to 27] | 3 [0 to 27]
Duration of ZDV during pregnancy - At Delivery [Median (Full Range); unit: weeks] | 10 [2 to 16] | 11 [5 to 18] | 10 [0 to 31] | 10 [0 to 31]
CD4 cell count at entry [Median (Full Range); unit: cells/uL] | 431 [262 to 1233] | 413 [251 to 1024] | 481 [262 to 1183] | 456 [251 to 1233]
CD4 cell count at delivery [Median (Full Range); unit: cells/uL] | 484 [70 to 1001] | 517 [198 to 1150] | 566 [222 to 1182] | 513 [70 to 1182]
Plasma HIV RNA at entry [Median (Full Range); unit: log10 copies/mL] | 3.48 [2.60 to 4.98] | 3.52 [1.00 to 4.99] | 3.54 [2.60 to 5.05] | 3.49 [1.00 to 5.05]
Plasma HIV-RNA at delivery [Median (Full Range); unit: log10 copies/mL] | 3.63 [1.70 to 4.90] | 3.36 [1.70 to 4.83] | 3.48 [1.70 to 4.71] | 3.48 [1.70 to 4.90]

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Women Who Develop One or More New NVP Resistance Mutations as Identified by Consensus Sequencing or Oligonucleotide Ligation Assay in Plasma (Sampling Was Done at Days 10,21,30, and Weeks 5,6, and 8 Postpartum).
Description: The incidence of new NVP resistance mutation in plasma HIV within 8 weeks postpartum in each randomized arm was estimated using an exact binomial confidence interval. If a resistance mutation was detected at any of the timepoints then an endpoint was met. Samples with VL <500 copies/mL were considered free of mutations. If a resistance result was missing for reasons other than VL <500 copies/ml (e.g.missed visit), it was conservatively imputed as resistant in the primary analysis.
Time Frame: within 8 weeks postpartum.
Population: All women who started treatment were included in an intention-to-treat analysis.
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- Arm A : LPV/r x 7d: NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, every 3 hours during labor and twice daily for 7 days postpartum ddI 250 mg orally (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 7 days postpartum, LPV/r 400/100mg orally twice daily at the onset of labor, during labor and for 7 days postpartum.
- Arm B : no LPV/r: NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, q3h during labor and twice daily for 30 days postpartum, ddI 250 mg orally (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 30 days postpartum.
- Arm C: LPV/r x 30d: NVP 200 mg orally, single dose at onset of labor,ZDV 300 mg orally at onset of labor, evry 3 hours during labor and twice daily for 30 days postpartum, ddI 250 mg orally (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 30 days postpartum, LPV/r 400/100mg orally twice daily at the onset of labor, during labor and for 30 days postpartum.
Arm/Group | Arm A : LPV/r x 7d | Arm B : no LPV/r | Arm C: LPV/r x 30d
Number analyzed (Participants) | 56 | 56 | 57
percent of participants | 7.1 [2.0 to 17.3] | 12.5 [5.2 to 24.1] | 5.3 [1.1 to 14.6]

2. Primary Outcome: The Proportion of Women in Each Randomized Arm Who Have One or More New NVP Resistance Mutations as Identified by Consensus Sequencing or Oligonucleotide Ligation Assay (OLA) in Plasma
Description: The incidence of new NVP resistance mutations at day 10 or week 6 postpartum in each randomized arm. Samples with viral load <500 copies/mL were considered free of mutations. If a resistance result was missing for reasons other than VL <500 copies/ml it was conservatively imputed as resistant in the primary analysis.
Time Frame: at Day 10 or Week 6 postpartum.
Population: All women who started treatment were included in an intention-to-treat analysis (according to randomized treatment assignment, regardless of compliance with the protocol)
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- Arm C : LPV/r x 30d: NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, every 3 hours during labor and twice daily for 30 days postpartum, ddI 250 mg orally (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 30 days postpartum, LPV/r 400/100mg orally twice daily at the onset of labor, during labor and for 30 days postpartum.
Arm/Group | Arm A : LPV/r x 7d | Arm B : no LPV/r | Arm C : LPV/r x 30d
Number analyzed (Participants) | 56 | 56 | 57
percent of participants | 3.6 [0.5 to 12.3] | 7.1 [2.0 to 17.3] | 5.3 [1.1 to 14.6]

3. Primary Outcome: Area Under the Curve Pharmacokinetic Outcome for LPV/r. (AUC ug*hr/mL)
Description: Data was analyzed with WinNonLin (Version 5.2, Pharsight, USA) using non-compartmental methods. The pharmacokinetic parameters were calculated using the linear-trapezoidal rule. Cpredose and C4hour at the two measurement times were compared within-subject using the Wilcoxon signed-rank test.
Time Frame: Within 72 hours postpartum and during the first 30 days postpartum
Population: 18 women were enrolled in this sub study,PK sampling was not performed in 2 women. Of the remaining 16 women, all completed the LPV/r PK sampling within 72 hours after delivery and at day 30 postpartum and had evaluable PK within 72 hours delivery but only 14 women had evaluable PK results at day 30 postpartum due to suspected poor drug adherence.
Measure: Median (Full Range); unit: ug*hr/mL
Groups:
- Within 72 Hrs Ppm; At Day 30 Ppm: ZDV, ddI, LPV/r x 30d
Arm/Group | Within 72 Hrs Ppm | At Day 30 Ppm
Number analyzed (Participants) | 16 | 14
ug*hr/mL | 99.7 [66.3 to 180.5] | NA [NA to NA] — Only 3 samples were collected at 30 days postpartum for PK assessment (pre-dose, 2 hours and 4 hours post-dose) and with these limited number of samples it was not possible to have a good estimate of the AUC and Cmax.
Statistical Analysis 1: Comparison: Within 72 Hrs Ppm vs At Day 30 Ppm; The null hypothesis was that there was no difference in within-subject Cpredose LPV/r plasma drug concentrations within 72 hours after delivery versus at 30 days postpartum; Test type: Superiority or Other; p = 0.009, wilcoxon Signed Rank Test — The p-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was two-sided P<0.05
Statistical Analysis 2: Comparison: Within 72 Hrs Ppm vs At Day 30 Ppm; The null hypothesis was that there was no difference in within-subject C4hour LPV/r plasma drug concentrations within 72 hours after delivery versus at 30 days postpartum; Test type: Superiority or Other; p = 0.048, Wilcoxon Signed Rank Test — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: The Proportion of Women in Each Randomized Arm Who Have One or More New NVP Resistance Mutations for the Subgroup of Women With Plasma HIV RNA >= 500 Copies/ml At Entry
Description: as for outcome 2
Time Frame: at Day 10 or Week 6 postpartum.
Population: Includes only the Subgroup of women with Plasma HIV RNA >= 500 copies/ml at Entry and who started treatment; analyzed using the intention-to-treat principle (according to assigned treatment, regardless of compliance with the protocol).
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- Arm A: LPV/r x 7d: NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, every 3 hours during labor and twice daily for 7 days postpartum, ddI 250 mg orally (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 7 days postpartum, LPV/r 400/100mg orally twice daily at the onset of labor, during labor and for 7days postpartum.
- Arm B: no LPV/r: NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, every 3 hours during labor and twice daily for 30 days postpartum, ddI 250 mg orally (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 30 days postpartum.
- Arm C : LPV/r x 30d: NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, q3h during labor and twice daily for 30 days postpartum, ddI 250 mg orally (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 30 days postpartum, LPV/r 400/100mg orally twice daily at the onset of labor, during labor and for 30 days postpartum.
Arm/Group | Arm A: LPV/r x 7d | Arm B: no LPV/r | Arm C : LPV/r x 30d
Number analyzed (Participants) | 41 | 42 | 43
percent of participants | 4.9 [0.6 to 16.6] | 9.5 [2.7 to 22.6] | 7.0 [1.5 to 19.1]

5. Secondary Outcome: The Proportion of Women With Any New ZDV, ddI, or LPV/r Resistance Mutations.
Time Frame: At Week 5 postpartum (ZDV) and at the first timepoint with viral load >=500 copies/ml after treatment discontinuation (ddI and LPV/r).
Population: All women who started treatment were included in an intention-to-treat analysis
Measure: Number; unit: percent of participants
Groups:
- Arm C: LPV/r x 30d: NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, every 3 hours during labor and twice daily for 30 days postpartum, ddI 250 mg orally (if body weight <60 kg) or 400 mg orally daily (if body weight >= 60 kg) at the onset of labor, during labor, and for 30 days postpartum, LPV/r 400/100mg orally twice daily at the onset of labor, during labor and for 30 days postpartum.
Arm/Group | Arm A : LPV/r x 7d | Arm B : no LPV/r | Arm C: LPV/r x 30d
Number analyzed (Participants) | 56 | 56 | 57
percent of participants
  The proportion of women with new ZDV resistance | 0 | 1.78 | 0
  The proportion of women with new ddI resistance | 0 | 0 | 0
  The proportion of women with new LPV/r resistance | 0 | 0 | 0

6. Secondary Outcome: Number of Women With Grade >=3 Events After Start of Study Treatment
Description: Adverse events were graded using the Division of AIDS (DAIDS) Table for Grading > the Severity of Adult and Pediatric Adverse Events (December 2004). All grade 3 and higher signs, symptoms, and laboratory toxicities (and events of any grade that led to a change in study treatment) were included.
Time Frame: After start of study Treatment (postpartum)
Population: All women who started treatment were included in an intention-to-treat analysis.
Measure: Number; unit: participants
Arm/Group | Arm A : LPV/r x 7d | Arm B : no LPV/r | Arm C: LPV/r x 30d
Number analyzed (Participants) | 56 | 56 | 57
participants | 2 | 0 | 2

7. Secondary Outcome: Proportion of Women With New NVP Resistance Mutation Within 8 Weeks Postpartum Who Had a NVP Resistance Mutation Detected at 72 Weeks Postpartum.
Description: Resistance mutations as identified by OLA in plasma samples or PBMC at 72 weeks postpartum amongst women who had new NVP resistance mutations within 8 weeks postpatrum. These results were based on the 13 women who developed a new NVP resistance mutation in the first 8 weeks postpartum. For the primary outcome measure 1, one particpant in arm A was unavailable for follow-up after week 5 and was conservatively imputed to have developed resistance mutation.
Time Frame: within 72 weeks postpartum
Population: amongst the participants who developed resistance within 8 weeks postpartum
Measure: Number; unit: participants
Arm/Group | Arm A : LPV/r x 7d | Arm B : no LPV/r | Arm C: LPV/r x 30d
Number analyzed (Participants) | 3 | 7 | 3
participants
  OLA in plasma samples | 0 | 0 | 0
  OLA in PBMC | 0 | 0 | 1

8. Secondary Outcome: Resistance Mutations in HIV Infected Infants
Description: Resistance mutations as identified by consensus sequencing or OLA
Time Frame: 24 weeks postpartum
Population: Amongst the infants who became HIV-infected.
Measure: Number; unit: participants
Arm/Group | Arm A : LPV/r x 7d | Arm B : no LPV/r | Arm C: LPV/r x 30d
Number analyzed (Participants) | 0 | 1 | 1
participants |  | 0 | 0

9. Secondary Outcome: Median HIV-1 Viral Load at 24 Weeks Postpartum in Women
Time Frame: at 24 weeks postpartum
Population: The number of particpants included in this analyses were for those for whom viral loads were available at 24 weeeks postpartum.
Measure: Median (Full Range); unit: log10 copies/mL
Groups:
- Arm A : LPV/r x 7d: NVP 200 mg orally, single dose at onset of labor, ZDV 300 mg orally at onset of labor, every 3 hours during labor and twice daily for 7 days postpartum, ddI 250 mg orally (if body weight <60 kg) or 400 mg orally QD (if body weight >= 60 kg) at the onset of labor, during labor, and for 7 days postpartum, LPV/r 400/100mg orally twice daily at the onset of labor, during labor and for 7 days postpartum.
Arm/Group | Arm A : LPV/r x 7d | Arm B : no LPV/r | Arm C: LPV/r x 30d
Number analyzed (Participants) | 54 | 55 | 54
log10 copies/mL | 4.3 [1.7 to 5.7] | 3.9 [1.7 to 5.3] | 4.0 [1.7 to 5.2]

10. Primary Outcome: Maximum Concentration Pharmacokinetic Outcome for LPV/r (Cmax ug/mL) .
Description: as for outcome 3
Time Frame: Within 72 hours postpartum and during the first 30 days postpartum
Population: as for outcome 3
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Within 72 Hrs Ppm | At Day 30 Ppm
Number analyzed (Participants) | 16 | 14
ug/mL | 11.2 [8.0 to 17.5] | NA [NA to NA] — Only 3 samples were collected at 30 days postpartum for PK assessment (pre-dose, 2 hours and 4 hours post-dose) and with these limited number of samples it was not possible to have a good estimate of the Cmax.

11. Primary Outcome: Pre-dose Concentration Pharmacokinetic Outcome for LPV/r (Cpredose ug/mL).
Description: as for outcome 3
Time Frame: Within 72 hours postpartum and during the first 30 days postpartum
Population: as for outcome 3
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Within 72 Hrs Ppm | At Day 30 Ppm
Number analyzed (Participants) | 16 | 14
ug/mL | 6.08 [2.34 to 13.64] | 9.17 [5.28 to 14.97]

12. Primary Outcome: Four (4) Hour Concentration Pharmacokinetic Outcome for LPV/r (C4hour ug/mL).
Description: as for outcome 3
Time Frame: Within 72 hours postpartum and during the first 30 days postpartum
Population: as for outcome 3
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Within 72 Hrs Ppm | At Day 30 Ppm
Number analyzed (Participants) | 16 | 14
ug/mL | 10.78 [8.01 to 16.72] | 12.96 [8.78 to 21.37]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were required to be reported for the entire duration for an individual subject i.e. from study enrollment until study completion or discontinuation of the subject from study participation for any reason.
Description: Expedited adverse event (EAE) reporting was at the DAIDS Intensive level: all deaths, congenital anomalies, fetal losses, or significant disabilities; also, suspected adverse drug reactions of grade >=3 for mothers or grade >=1 for infants (grade 1=mild, 2=moderate, 3=severe, 4=life threatening, 5=death per the 12/2--4 DAIDS AE Grading Table).
Groups:
- Mother: LPV/r x 7d; Infant: LPV/r x 7d: NVP 200 mg orally, single dose at onset
- Mother: no LPV/r; Infant: no LPV/r: ZDV & ddI x 30d
- Mother: LPV/r x 30d; Infant: LPV/r x 30d: ZDV, ddI, LPV/r x 30d
Arm/Group | Mother: LPV/r x 7d | Mother: no LPV/r | Mother: LPV/r x 30d | Infant: LPV/r x 7d | Infant: no LPV/r | Infant: LPV/r x 30d
Serious Adverse Events (participants affected / at risk) | 0/56 | 1/56 | 2/57 | 34/56 | 32/57 | 33/57
Other Adverse Events (participants affected / at risk) | 33/56 | 43/56 | 45/57 | 48/56 | 51/57 | 49/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mother: LPV/r x 7d (N=56) | Mother: no LPV/r (N=56) | Mother: LPV/r x 30d (N=57) | Infant: LPV/r x 7d (N=56) | Infant: no LPV/r (N=57) | Infant: LPV/r x 30d (N=57)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 17 | 8 | 10
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 4 | 1
Neutropenia neonatal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1 | 1
ABO haemolytic disease of newborn (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Congenital hypothyroidism (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fallot's tetralogy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Trisomy 21 (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 10 | 11 | 10
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 3 | 6 | 2
Blood calcium increased (Investigations) | 0 | 0 | 0 | 5 | 1 | 4
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 2 | 6
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 4 | 2 | 2
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2
Blood sodium increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 3 | 0 | 2
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4 | 2
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 1
Neonatal hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 2
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 1 | 2
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mother: LPV/r x 7d (N=56) | Mother: no LPV/r (N=56) | Mother: LPV/r x 30d (N=57) | Infant: LPV/r x 7d (N=56) | Infant: no LPV/r (N=57) | Infant: LPV/r x 30d (N=57)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 11 | 15 | 12
Anaemia neonatal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 4 | 0 | 3
Ear pain (Ear and labyrinth disorders) | 3 | 2 | 0 | 0 | 0 | 0
Conjunctival discolouration (Eye disorders) | 0 | 0 | 0 | 5 | 1 | 4
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 3
Eye discharge (Eye disorders) | 1 | 0 | 0 | 2 | 3 | 6
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 2 | 5 | 3 | 4
Diarrhoea neonatal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4 | 2 | 0 | 1 | 1
Pyrexia (General disorders) | 6 | 9 | 8 | 9 | 10 | 16
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 4 | 3
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 8 | 6 | 11
ABO incompatibility (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 3
Bronchitis (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 5 | 6 | 2 | 5 | 7
Pharyngitis (Infections and infestations) | 1 | 4 | 2 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 6 | 3 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 2 | 4 | 1 | 2
Vulvovaginal candidiasis (Infections and infestations) | 2 | 2 | 4 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 5 | 1 | 1 | 2 | 5
Aspartate aminotransferase increased (Investigations) | 4 | 7 | 5 | 6 | 4 | 3
Blood bicarbonate abnormal (Investigations) | 0 | 0 | 0 | 6 | 7 | 3
Blood bilirubin increased (Investigations) | 2 | 1 | 3 | 1 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 5
Blood glucose abnormal (Investigations) | 3 | 4 | 2 | 2 | 6 | 3
Blood glucose decreased (Investigations) | 6 | 3 | 3 | 0 | 2 | 2
Blood glucose increased (Investigations) | 8 | 3 | 7 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 5 | 4 | 6
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 7 | 7 | 6
Cardiac murmur (Investigations) | 0 | 0 | 0 | 4 | 1 | 3
Haemoglobin abnormal (Investigations) | 1 | 0 | 2 | 23 | 15 | 20
Haemoglobin decreased (Investigations) | 15 | 16 | 21 | 22 | 18 | 22
Neutrophil count decreased (Investigations) | 1 | 2 | 4 | 5 | 8 | 3
Platelet count decreased (Investigations) | 4 | 2 | 2 | 3 | 0 | 2
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 2 | 0
Hypothermia neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 3 | 0 | 3
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 14 | 12 | 15
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 3 | 1 | 0
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 3 | 3
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 2 | 6 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 3 | 3 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 3 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 3 | 7 | 5 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 1 | 1
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 2 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 3 | 8 | 5 | 11
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 4 | 4 | 3 | 2 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 4 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 5 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5 | 1 | 1
Pallor (Vascular disorders) | 0 | 0 | 0 | 4 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights".